CLINICAL TRIAL: NCT02367092
Title: Exercise Intervention in Liver Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Johns Hopkins University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-14783
Record Dates: First submitted 2014-12-20; First posted 2015-02-20 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: End Stage Liver Disease; Sarcopenia; Liver Cirrhoses
Keywords: Liver Transplantation
MeSH Terms: conditions — End Stage Liver Disease; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Program (Experimental): The exercise intervention consists of a 30 minute exercise session led by an instructor through a DVD or a video available on the internet.
  Interventions: Behavioral: Exercise Program
- Standard of care (No Intervention): Standard of care which consists of encouragement to exercise by the subject's transplant clinician.

INTERVENTIONS:
Behavioral: Exercise Program — They will perform low-intensity, low-resistance exercise facilitated by a DVD video in their home. This exercise program lasts for 30 minutes at a time. Patients will be instructed to engage in this exercise program 3-4 times per week but not more often than 4 times per week. Pre-transplant patients will be asked to do the exercises from enrollment to transplant. Post-transplant patients will be asked to do the exercises for 6 months.
  Arms: Exercise Program

SUMMARY:
The purpose of this study is to learn more about the effects of exercise on functional status and outcomes on patients with end-stage liver disease on the liver transplant waiting list and who have undergone liver transplantation.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a home-based exercise intervention on outcomes in liver transplant candidates and recipients. This home-based intervention consists of a 30-minute exercise session available on digital video disc or on the internet. This intervention was originally developed to improve functional status in community-dwelling older adults and therefore, has been designed to maximize the safety for even the most frail individuals. Subjects enrolled in this study will be randomized to one of two arms: (a) the exercise intervention arm in which the subjects will be asked perform this exercise session three to four times per week or (b) the standard-of-care arm in which the patient will be encouraged to exercise by their transplant clinician at every clinic visit. Subjects in the exercise intervention arm will undergo this intervention for 6 months. All subjects will be followed for up to two years from the time of enrollment to ascertain outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>=18 years of age)
* Listed for liver transplantation or post-liver transplantation
* English speaking

Exclusion Criteria:

* Contraindications to weight-bearing exercise
* Non-English speaking
* Requires an assistive device for ambulation
* Active hepatic encephalopathy at the time of baseline assessment for enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-07; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Liver Frailty Index | 12 and 24 weeks after enrollment
  Liver Frailty Index as measured by score in functional assessments of grip strength (kg), balance (seconds), and chair stands (seconds).

SECONDARY OUTCOMES:
Mortality at 24 weeks | 1 year
  Mortality status at 24 weeks
Hospitalized days at 24 weeks | 1 year
  Number of days in the hospital from baseline to 24 weeks
Quality of Life by CLDQ | 12 and 24 weeks after enrollment
  Quality of life assessed by the CLDQ at 12 and 24 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Lai, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina

REFERENCES:
- [Background] Murray KF, Carithers RL Jr; AASLD. AASLD practice guidelines: Evaluation of the patient for liver transplantation. Hepatology. 2005 Jun;41(6):1407-32. doi: 10.1002/hep.20704. No abstract available. PMID 15880505
- [Background] Lai JC, Feng S, Terrault NA, Lizaola B, Hayssen H, Covinsky K. Frailty predicts waitlist mortality in liver transplant candidates. Am J Transplant. 2014 Aug;14(8):1870-9. doi: 10.1111/ajt.12762. Epub 2014 Jun 16. PMID 24935609
- [Background] Dasarathy S. Consilience in sarcopenia of cirrhosis. J Cachexia Sarcopenia Muscle. 2012 Dec;3(4):225-37. doi: 10.1007/s13539-012-0069-3. Epub 2012 May 31. PMID 22648736
- [Background] Jones JC, Coombes JS, Macdonald GA. Exercise capacity and muscle strength in patients with cirrhosis. Liver Transpl. 2012 Feb;18(2):146-51. doi: 10.1002/lt.22472. PMID 22139897
- See also: United Network for Organ Sharing — https://optn.transplant.hrsa.gov